CLINICAL TRIAL: NCT02406534
Title: A Prospective, Observational Study of COPD Patients in U.S. Hospitals
Status: Withdrawn | Type: Observational
Why Stopped: Study entered in error
Sponsor: EPI-Q (Other)
Responsible Party: Sponsor
Other Study IDs: 000
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Pulmonary Function
  Interventions: Behavioral: HRQoL surveys
- Reduced Pulmonary Function
  Interventions: Behavioral: HRQoL surveys

INTERVENTIONS:
Behavioral: HRQoL surveys

SUMMARY:
This is an observational study to evaluate the relationship between pulmonary function and the patient reported health-related quality of life (HRQoL) and chronic obstructive pulmonary disease (COPD) related admissions. Patients with COPD will be approached to participate in the study. Pulmonary function will be measured on consented, eligible patients. The pulmonary function measurement collected will be used for cohort assignment. The prospective follow up period will monitor the cohorts for evidence of readmission and to assess HRQoL.

ELIGIBILITY:
Inclusion Criteria:

≥ 18 years of age Fluent in English Current hospital admission is for COPD Diagnosis of COPD for at least 1 year prior to enrollment

Exclusion Criteria:

Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COPD patients admitted for a COPD exacerbation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
COPD related readmissions | 6 months
Health related quality of life (HRQoL) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Caroselli, Study Director — EPI-Q